CLINICAL TRIAL: NCT03138694
Title: Adnexal Mass After Methotrexate Treatment for Ectopic Pregnancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 614-16-TLV
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Ectopic Pregnancies
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methotrexate injection: Patients with Ectopic pregnancy treated with Methotrexate injection.
  Interventions: Other: BHCG monitoring
- Self resolution: Patients with Ectopic pregnancy that had signs of self resolution with our "Watchful waiting" protocol.
  Interventions: Other: BHCG monitoring

INTERVENTIONS:
Other: BHCG monitoring — Participants in the study will be invited to our outpatient clinic for BHCG monitoring including blood count and BHCG levels test and serial Transvaginal Ultrasound examination

SUMMARY:
Ectopic pregnancies are a common morbidity in the gynaecological field. Previous work done by our team has shown the benefits of conservative treatment with only BHCG (Beta-Human Chorionic Gonadotropin) monitoring, proving that a vast number of patients will have a self resolution without the need for any further medical intervention. In addition, our working hypothesis is that this process in contrast to Methotrexate is a more physiologic one with less inflammatory and necrosis reaction.

OBJECTIVE To measure and compare the size of the ectopic mass and monitor BHCG levels of women treated with Methotrexate and those that had a self resolution process of their ectopic pregnancy.

Investigators aim to prove that the mass will have an enlargement trend after Methotrexate in contrast to being stable or decrease in size with conservative treatment.

DETAILED DESCRIPTION:
Ectopic pregnancies are a common morbidity in the gynaecological field. Previous work done by our team has shown the benefits of conservative treatment with only BHCG (Beta-Human Chorionic Gonadotropin) monitoring, proving that a vast number of patients will have a self resolution without the need for any further medical intervention. In addition, our working hypothesis is that this process in contrast to Methotrexate is a more physiologic one with less inflammatory and necrosis reaction.

OBJECTIVE To measure and compare the size of the ectopic mass and monitor BHCG levels of women treated with Methotrexate and those that had a self resolution process of their ectopic pregnancy.

Investigators aim to prove that the mass will have an enlargement trend after Methotrexate in contrast to being stable or decrease in size with conservative treatment.

PATIENTS & METHODS Patients that will be offered to join the study are those that will be with either treated by a Methotrexate injection or those that had signs of self resolution with our "Watchful waiting" protocol.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted and treated for a diagnosis of Ectopic pregnancy in The Department of Gynecology, Lis Maternity Hospital.

Exclusion Criteria:

none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted and treated for a diagnosis of Ectopic pregnancy in The Department of Gynecology, Lis Maternity Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
ectopic mass size | up to 6 weeks.
  measuring and comparing the size of the ectopic mass

SECONDARY OUTCOMES:
BHCG values | up to 6 weeks.
  BHCG levels test in blood

CONTACTS AND LOCATIONS:
Overall Officials: Ishai Levin, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No